CLINICAL TRIAL: NCT00298441
Title: Effect of IVIR Frequency on Anemia Correction and Oxidative Stress Formation and in Hemodialysis Patients
Brief Title: Efficacy of Intravenous Iron Administration in Hemodialysis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kumamoto University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KU-Neph-05-001
Record Dates: First submitted 2006-02-28; First posted 2006-03-02 (Estimated); Last update posted 2008-05-12 (Estimated); Status verified 2008-05

CONDITIONS: Chronic Renal Failure; Hemodialysis; Renal Anemia; Iron Deficiency Anemia
Keywords: intravenous iron administration
MeSH Terms: conditions — Kidney Failure, Chronic; Anemia, Iron-Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: chondroitin sulfate-iron colloid

SUMMARY:
The purpose of this study is to determine whether the frequency of intravenous iron administration has an effect on anemia correction and oxidative stress formation in hemodialysis patients.

DETAILED DESCRIPTION:
In patients who are on chronic hemodialysis (HD), anemia is a major complication and is associated with poor clinical outcomes. Consequently, management of anemia by recombinant erythropoietin is reported consistently to improve outcome measures in HD patients. Because iron is essential for hemoglobin formation, as is erythropoietin, most patients routinely receive iron intravenously (IVIR) for anemia correction. Although IVIR has been shown to improve both survival and quality of life of HD patients, it has been suggested that IVIR may enhance the generation of hydroxyl radicals in the body through the inflammation process and the Fenton reaction. Previously we demonstrated that that serum albumin is highly oxidized in HD patients and that IVIR on these patients significantly increased the oxidation status of albumin.

In 2004, the committee on the guidelines of the Japanese Society for Dialysis Therapy (JSDT) published the original Japanese "Guidelines for Renal Anemia in Chronic Hemodialysis Patients". In the JSDT guidelines 2004, the committee recommended two IVIR schedules for iron deficient patients; 1) administer 40 mg of IV iron at the end of dialysis session 3 times a week for 4 weeks (total 520 mg of iron), 2) administer 40 mg of IV iron at the end of dialysis session once a week for 3 months (total 520 mg of iron). Both administration schedules are effective for the correction of iron deficiency and consequently for the amelioration of anemia. However, the effect of IVIR frequency (three times a week vs. once a week) on the oxidative stress formation has not been investigated before.

Comparison: the two IVIR schedules recommended by the JSDT guideline 2004 will be compared by measuring both hemoglobin and oxidized albumin in chronic HD patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of chronic renal failure
* Clinical diagnosis of iron deficiency anemia
* Must be on regular hemodialysis

Exclusion Criteria:

* Allergic to intravenous iron administration

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2005-06; Primary Completion 2006-05 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
hemoglobin levels at 24 weeks
oxidized albumin levels at 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kenichiro Kitamura, M.D., Ph.D., Principal Investigator — Kumamoto University
Locations (2):
- Japan (2):
  - Midorigaoka Clinic, Arao, Kumamoto
  - Kumamoto University Hospital, Kumamoto, Kumamoto

REFERENCES:
- [Background] Anraku M, Kitamura K, Shinohara A, Adachi M, Suenga A, Maruyama T, Miyanaka K, Miyoshi T, Shiraishi N, Nonoguchi H, Otagiri M, Tomita K. Intravenous iron administration induces oxidation of serum albumin in hemodialysis patients. Kidney Int. 2004 Aug;66(2):841-8. doi: 10.1111/j.1523-1755.2004.00813.x. PMID 15253741